CLINICAL TRIAL: NCT06385418
Title: Fluorouracil Treatment Via Colon for Colorectal Cancer: an Exploratory Study
Brief Title: Fluorouracil Treatment Via Colon for Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Vice President, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WST-CRC-202404
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer
Keywords: Fluorouracil; Transendoscopic enteral tubing; Thermosensitive hydrogel; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Colonic local administration of fluorouracil with enhanced adhesion (Experimental): Fluorouracil is administered via the colon as an injectable solution at a dose of 500 mg per day for 6 days, along with poloxamer 407 and poloxamer 188 used as thermosensitive hydrogel to enhance adhesion.
  Interventions: Drug: Colonic local administration of fluorouracil with enhanced adhesion

INTERVENTIONS:
Drug: Colonic local administration of fluorouracil with enhanced adhesion — Fluorouracil is administered via the colon as an injectable solution at a dose of 500 mg per day for 6 days, along with poloxamer 407 and poloxamer 188 used as thermosensitive hydrogel to enhance adhesion.

SUMMARY:
Fluorouracil (5-FU) is a commonly used drug for colorectal cancer (CRC). Thermosensitive hydrogel presents a promising carrier for 5-FU to address challenges encountered with traditional administration methods. We propose an integrated approach utilizing colonic transendoscopic enteral tubing to cover the entire colon flexibly, coupled with a thermo-sensitive gel to enhance the adhesion of 5-FU. This clinical trial aims to assess the feasibility, safety, and efficacy of this approach for treating CRC.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese individuals aged 18 to 75 years, both male and female;
2. Histologically confirmed diagnosis of colorectal cancer with measurable primary lesion according to RECIST 1.1;
3. ECOG performance status ≤2;
4. Expected survival of more than 3 months;
5. Multidisciplinary team consensus that the patient is suitable for adding local chemotherapy to the established tumor treatment regimen;
6. Adequate organ function meeting the following criteria: (1) Absolute neutrophil count ≥1.5 × 10^9/L, platelets ≥100 × 10^9/L, hemoglobin ≥90 g/L; (2) Total bilirubin ≤1.5 times the upper limit of normal (patients with biliary drainage via retrograde techniques included); ALT and AST ≤5 times the upper limit of normal, and for patients with liver metastases, serum total bilirubin less than or equal to 3 times the upper limit of the normal reference range; (3) Creatinine <120 μmol/L, or MDRD estimated glomerular filtration rate >60 mL/min; (4) Doppler echocardiography assessment: Left ventricular ejection fraction (LVEF) ≥50%;
7. Women of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days before enrollment, and sexually active men or women agree to use appropriate contraception during the trial and for 8 weeks after the last dose of investigational drug;
8. Suitable physical condition and personal willingness to undergo colonic transendoscopic enteral tubing;
9. Willingness to cooperate with physicians, and agree to regular follow-up visits and examinations as recommended after completion of treatment;
10. Agreement to specimen collection and voluntary signing of a written informed consent form.

Exclusion Criteria:

1. Uncontrolled cardiovascular diseases, such as congestive heart failure (NYHA III-IV), coronary artery disease, cardiomyopathy, arrhythmias, or hemodynamic instability at enrollment, with a risk of significant events during the treatment period;
2. Active severe clinical infections (≥ Grade 2 according to NCI-CTCAE version 5.0), including fungal, viral, or tuberculosis infections within the gastrointestinal tract;
3. Coagulation abnormalities with bleeding tendencies (who do not meet the criteria of having a normal INR without the use of anticoagulants within 14 days prior to enrollment). Participants receiving anticoagulants or vitamin K antagonists such as warfarin or heparin are excluded unless their international normalized ratio (INR) is ≤1.5, with allowance for low-dose warfarin (1 mg orally once daily) or low-dose aspirin (daily dose not exceeding 100 mg) for prophylaxis;
4. History of immunodeficiency or other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
5. Known progressive or actively treated other malignancies requiring intervention, except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ;
6. Presence of other serious diseases that would render the subject ineligible for enrollment as determined by the investigator;
7. Breastfeeding women;
8. Known allergy or intolerance to the investigational drug or its excipients;
9. Participation in another drug clinical trial within the past four weeks;
10. Lack of legal capacity or restricted legal capacity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (according to RECIST1.1, investigator assessment) | One, three, and six months (or until conversion to surgery) after the initial treatment
  Objective response rate (ORR) is defined as complete response (CR) and partial response (PR) proportion of participants.

SECONDARY OUTCOMES:
Progression-free survival | One, three, and six months (or until conversion to surgery) after the initial treatment
  Progression-free survival (PFS) is defined as the time from the first initiation of study regimen treatment to the first imaging disease progression or the time of death, whichever occurs first.
Overall survival | Every 3 months up to 24 months after the end of treatment
  Overall survival (OS) is defined as the time from the first initiation of the study regimen to death from any cause time.
Disease control rate (according to RECIST1.1, investigator assessment) | One, three, and six months (or before conversion to surgery) after the initial treatment
  Disease control rate (DCR) is defined as the proportion of participants with complete response (CR), partial response (PR) and stable disease (SD) × 100%.
Drop period to ensure operation resection | Time from the first treatment to 4-6 cycles (each cycle is 28 days) of treatment
  Drop period to ensure operation resection is defined as the proportion of participants whose tumors shrink following study induction therapy, thereby enhancing the safety and feasibility of surgical removal.
Converted resection rate | Time from the first treatment to 4-6 cycles (each cycle is 28 days) of treatment
  Surgical conversion rate, defined as the proportion of participants who achieved gross complete resection after 4-6 courses of study induction therapy.
Actual R0 resection rate | Time from the first treatment to 4-6 cycles (each cycle is 28 days) of treatment
  Actual R0 resection rate is defined as the proportion of participants who achieved R0 surgical resection after 4-6 courses of study induction therapy.
The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | Throughout the treatment period and continuing for an additional 6 months after the treatment concludes, an average of 1 year
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD, PhD, Principal Investigator — Department of Microbiota Medicine & Medical Center for Digestive Diseases
Locations (1):
- The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Sun W, Zhang N, Li A, Zou W, Xu W. Preparation and evaluation of N(3)-O-toluyl-fluorouracil-loaded liposomes. Int J Pharm. 2008 Apr 2;353(1-2):243-50. doi: 10.1016/j.ijpharm.2007.11.017. Epub 2007 Nov 17. PMID 18155370
- [Background] Longley DB, Harkin DP, Johnston PG. 5-fluorouracil: mechanisms of action and clinical strategies. Nat Rev Cancer. 2003 May;3(5):330-8. doi: 10.1038/nrc1074. PMID 12724731
- [Background] Liu G, Franssen E, Fitch MI, Warner E. Patient preferences for oral versus intravenous palliative chemotherapy. J Clin Oncol. 1997 Jan;15(1):110-5. doi: 10.1200/JCO.1997.15.1.110. PMID 8996131
- [Background] Galandiuk S, Wrightson W, Marr L, Myers S, LaRocca RV. Suppository delivery of 5-fluorouracil in rectal cancer. Ann Surg Oncol. 1996 May;3(3):270-6. doi: 10.1007/BF02306282. PMID 8726182
- [Background] Kulkarni R, Fanse S, Burgess DJ. Mucoadhesive drug delivery systems: a promising noninvasive approach to bioavailability enhancement. Part II: formulation considerations. Expert Opin Drug Deliv. 2023 Mar;20(3):413-434. doi: 10.1080/17425247.2023.2181332. Epub 2023 Feb 22. PMID 36803264
- [Background] Zarrintaj P, Ramsey JD, Samadi A, Atoufi Z, Yazdi MK, Ganjali MR, Amirabad LM, Zangene E, Farokhi M, Formela K, Saeb MR, Mozafari M, Thomas S. Poloxamer: A versatile tri-block copolymer for biomedical applications. Acta Biomater. 2020 Jul 1;110:37-67. doi: 10.1016/j.actbio.2020.04.028. Epub 2020 May 15. PMID 32417265
- [Background] Al Sabbagh C, Seguin J, Agapova E, Kramerich D, Boudy V, Mignet N. Thermosensitive hydrogels for local delivery of 5-fluorouracil as neoadjuvant or adjuvant therapy in colorectal cancer. Eur J Pharm Biopharm. 2020 Dec;157:154-164. doi: 10.1016/j.ejpb.2020.10.011. Epub 2020 Oct 22. PMID 33222768
- [Background] Seguin J, Pimpie C, Roy P, Al Sabbagh C, Pocard M, Mignet N, Boudy V. Combination of tumor cell anti-adhesion and anti-tumor effect to prevent recurrence after cytoreductive surgery in a mice model. Eur J Pharm Biopharm. 2021 Dec;169:37-43. doi: 10.1016/j.ejpb.2021.01.020. Epub 2021 Mar 14. PMID 33727143
- [Background] Zhang F, Lu G, Wang X, Wu L, Li R, Nie Y. Concept, breakthrough, and future of colonic transendoscopic enteral tubing. Chin Med J (Engl). 2024 Mar 20;137(6):633-635. doi: 10.1097/CM9.0000000000003020. Epub 2024 Feb 7. No abstract available. PMID 38321613